CLINICAL TRIAL: NCT01621464
Title: Closed Loop Stimulation for Neuromediated Syncope
Brief Title: Closed Loop Stimulation for Neuromediated Syncope (SPAIN Study)
Acronym: SPAIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spanish Society of Cardiology (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Principal Investigator, Gonzalo Barón-Esquivias, MD, PhD, FESC, member of Syncope Working Group (within Section of Electrophysiology and Arrhythmias), Spanish Society of Cardiology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SPAIN
Record Dates: First submitted 2012-06-11; First posted 2012-06-18 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Syncope, Vasovagal
Keywords: Neuromediated syncope; Tilt test; Pacemaker; CLS sensor
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Pacemaker implanted but NO pacing (mode DDI, 30 bpm and sub-threshold)
  Interventions: Device: Pacemaker with Closed Loop Stimulation (CLS sensor)
- CLS group (Experimental): pacemaker implanted programmed with the contractility sensor activated (mode DDD-CLS)
  Interventions: Device: Pacemaker with Closed Loop Stimulation (CLS sensor)

INTERVENTIONS:
Device: Pacemaker with Closed Loop Stimulation (CLS sensor) — Crossover: 1 year at control group and 1 year at CLS group (randomized which group goes first)
  Other Names: BIOTRONIK; Neuromediated Syncope

SUMMARY:
Physiological stimulation therapy effectiveness will be proved with contractility sensor or CLS sensor (Closed Loop Stimulation), in BIOTRONIK CLS pacemakers to prevent from neuromediated syncope. Furthermore, not only will be investigated if this system eradicates syncopes, but also if the number of presyncopal episodes is reduced.

ELIGIBILITY:
Inclusion Criteria:

* Patients that fulfill the requirements of the study:

  * Patients with 5 previous neuromediated syncopes
  * Positive Tilt test, Cardioinhibitory response, heart rate < 40 bpm for at least 10'' or pauses > 3''
  * Patient ≥ 40 years
  * No cardiopathy present
* Patients without the following contraindications:

  * Drug treatment with β-blockers
  * Chronic Polyneuropathy
  * All contraindications for DDD or DDDR pacing (as per clinical guidelines SEC, 2002)
* Geographically stable patients and able to attend all follow ups
* Patients that have signed the informed consent

Exclusion Criteria:

* Patients that do NOT fulfill the inclusion criteria mentioned above
* Patients with the contraindications indicated above
* Patients with syncopes due to Carotid Sinus Hypersensitivity
* Other syncope causes different to the CNS
* Patients involved in other clinical studies
* Pregnant women or in age bearing that are not using at least 2 contraception methods

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2006-05; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of number of syncopes | 1 year
  Demonstrate that pacing therapy regulated by an inotropic sensor (CLS) is effective for the suppression of the neuromediated syncope

SECONDARY OUTCOMES:
Time reduction to the first syncope | 1 year
  Time reduction to 1st syncope: Time from the implantation to the 1st recurrence of the syncope.
Reduction of the recurrence of presyncopal symptoms | 1 year
  Reduction of the recurrence of presyncopal symptoms: Since the CLS sensor can detect any changes in contractility, and presyncopal symptoms are preceded by a contractility increase, it is thought that CLS group patients will suffer less from these symptoms.
Improvement of Quality of Life | 1 year
  Improvement of Quality of Life: Syncope produces uncertainties and fear to the patients. This will be checked if pacemaker implant improves QOL of these patients and if a specific programming scheme influences the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Barón Esquivias, MD PhD FESC, Principal Investigator — Spanish Society of Cardiology
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Sevilla, Spain

REFERENCES:
- [Derived] Baron-Esquivias G, Moya-Mitjans A, Martinez-Alday J, Ruiz-Granell R, Lacunza-Ruiz J, Garcia-Civera R, Gutierrez-Carretero E, Romero-Garrido R, Morillo CA. Impact of dual-chamber pacing with closed loop stimulation on quality of life in patients with recurrent reflex vasovagal syncope: results of the SPAIN study. Europace. 2020 Feb 1;22(2):314-319. doi: 10.1093/europace/euz294. PMID 31713631
- [Derived] Baron-Esquivias G, Morillo CA, Moya-Mitjans A, Martinez-Alday J, Ruiz-Granell R, Lacunza-Ruiz J, Garcia-Civera R, Gutierrez-Carretero E, Romero-Garrido R. Dual-Chamber Pacing With Closed Loop Stimulation in Recurrent Reflex Vasovagal Syncope: The SPAIN Study. J Am Coll Cardiol. 2017 Oct 3;70(14):1720-1728. doi: 10.1016/j.jacc.2017.08.026. PMID 28958328